CLINICAL TRIAL: NCT02887391
Title: Comparing Nutritional Status of In-centre Nocturnal Hemodialysis Patients to Conventional Hemodialysis Patients: A Prospective Cohort Study
Brief Title: Comparing Nutritional Status of In-centre Nocturnal Hemodialysis Patients to Conventional Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Associate Professor Medicine, University of Calgary
Other Study IDs: E-2358
Record Dates: First submitted 2016-08-15; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: hemodialysis; nutritional status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conventional Hemodialysis: Control group 4 hours of hemodialysis 3x per week (12 hours hemodialysis/week)
  Interventions: Other: No intervention - observational study
- In-Centre Nocturnal Hemodialysis: 8 hours of hemodialysis 3x per week (24 hours hemodialysis/week)
  Interventions: Other: No intervention - observational study

INTERVENTIONS:
Other: No intervention - observational study — No intervention - observational study

SUMMARY:
Although hemodialysis is life-saving, unfortunately, people on dialysis often have declining health, quality of life as well as poor nutritional status. Hemodialysis patients must follow a very restrictive diet, and many patients do not eat well and usually report poor appetites. A new approach to dialysis is being used in some hospitals in Alberta and elsewhere, called in-centre nocturnal hemodialysis. This in-centre nocturnal dialysis allows people to receive their dialysis at a hospital or clinic while they sleep. Since this in-centre nocturnal dialysis gives people 8-hour hemodialysis treatment 3 times per week (24 hours of dialysis per week) the patients have better removal of the waste products from their bodies than conventional hemodialysis (an average of 12 hours per week). Also of importance, when using in-centre nocturnal dialysis, people will have more time during the day to work, spend with family, as well as have time to shop for food, to cook and even to eat, which in turn will likely result in improvement in the quality of their lives. This study will follow 10 patients on conventional dialysis and 10 patients on in-centre nocturnal dialysis for 6 months and compare their food intake, muscle mass, weight, body mass index (BMI) and nutrition-related lab tests. The purpose of this study is to determine whether there is an improvement in the nutritional status of the in-centre nocturnal hemodialysis patients compared to the nutritional status of conventional hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* referred to the in-centre nocturnal hemodialysis program
* medically stable
* undergo hemodialysis three to four times per week for a minimum of three hours per week
* able to provide written, informed consent

Exclusion Criteria:

* younger than 18 years old
* have a current diagnosis with palliative status (e.g. cancer) or have active disease
* have had a prolonged hospitalization (>3 weeks) within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at all hemodialysis (HD) sites in the Southern Alberta Renal Program may be included. These sites include: Foothills Medical Center HD, Northland HD, Fanning HD, Sheldon Chumir HD, South Calgary HD, Peter Lougheed HD, and Sunridge HD in Calgary, AB.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Malnutrition Inflammation Score (MIS) | Baseline & 6 months
  A survey/tool that uses both subjective global assessment and objective laboratory measures to evaluate nutritional status. Change from baseline MIS at 6 months will be measured in both groups.

SECONDARY OUTCOMES:
Quality of Life | Baseline & 6 months
  KDQOL (SF-36) will be used to measure the quality of life in both groups at baseline and change after 6 months.
Dietary Intake | Baseline & 6 months
  3 day food records will be administered to document changes in dietary intake. Will be measured at baseline and change after 6 months in both groups.
Appetite | Baseline & 6 months
  Simplified Nutritional Appetite Questionnaire (SNAQ) will be administered to document changes in appetite. Will be measured at baseline and change after 6 months in both groups.
Interdialytic Weight Gain | Baseline & 6 months
  Measurement of fluid weight gain between dialysis sessions; Will be measured in both groups at baseline and after 6 months.
Body Mass Index (BMI) | Baseline & 6 months
  Body Mass Index (BMI) will be used to assess change in weight over time. Will be measured in both groups at baseline and after 6 months.
Triceps Skinfold Thickness | Baseline & 6 months
  Triceps skinfold thickness will be used to assess changes in muscle and fat mass over time. Will be measured in both groups at baseline and after 6 months.
Mid Arm (Muscle) Circumference | Baseline & 6 months
  Mid arm (muscle) circumference will be used to assess changes in muscle and fat mass over time. Will be measured in both groups at baseline and after 6 months.
Handgrip Strength | Baseline & 6 months
  Handgrip strength will be used to assess changes in muscle strength over time. Will be measured in both groups at baseline and after 6 months.
Bio-electrical Impedance | Baseline & 6 months
  This is completed as one measurement to assess body composition (fat, fluid, muscle). Will be measured at baseline and after 6 months in both groups.
Serum Albumin | Baseline & 6 months
  Serum albumin will be measured as part of hemodialysis standard of care. Change in baseline serum albumin will be evaluated at 6 months.
C-reactive protein (CRP) | Baseline & 6 months
  C-reactive protein will be measured as part of hemodialysis standard of care. Change in baseline CRP will be evaluated at 6 months.
Total iron binding capacity (TIBC) | Baseline & 6 months
  Total iron binding capacity (TIBC) will be measured as part of hemodialysis standard of care. Change in baseline TIBC will be evaluated at 6 months.
Phosphate Binders | Baseline & 6 months
  Changes in use and number/dose of phosphate binders will be measured at baseline and after 6 months in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer MacRae, MSc, MD, Principal Investigator — University of Calgary; Tanis Fenton, PhD, RD, Principal Investigator — University of Calgary; Rebecca Holmes, BCom, BSc, Study Director — University of Calgary
Locations (1):
- Alberta Health Services Southern Alberta Renal Program, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared

REFERENCES:
- [Background] Lacson E Jr, Xu J, Suri RS, Nesrallah G, Lindsay R, Garg AX, Lester K, Ofsthun N, Lazarus M, Hakim RM. Survival with three-times weekly in-center nocturnal versus conventional hemodialysis. J Am Soc Nephrol. 2012 Apr;23(4):687-95. doi: 10.1681/ASN.2011070674. Epub 2012 Feb 23. PMID 22362905
- [Background] Lacson E Jr, Wang W, Lester K, Ofsthun N, Lazarus JM, Hakim RM. Outcomes associated with in-center nocturnal hemodialysis from a large multicenter program. Clin J Am Soc Nephrol. 2010 Feb;5(2):220-6. doi: 10.2215/CJN.06070809. Epub 2009 Dec 3. PMID 19965529
- [Background] Demirci C, Ozkahya M, Demirci MS, Asci G, Kose T, Colak T, Duman S, Toz H, Ergin P, Adam SM, Ok E. Effects of three times weekly eight-hour nocturnal hemodialysis on volume and nutritional status. Am J Nephrol. 2013;37(6):559-67. doi: 10.1159/000351182. Epub 2013 May 30. PMID 23735837
- [Background] Ikizler TA, Cano NJ, Franch H, Fouque D, Himmelfarb J, Kalantar-Zadeh K, Kuhlmann MK, Stenvinkel P, TerWee P, Teta D, Wang AY, Wanner C; International Society of Renal Nutrition and Metabolism. Prevention and treatment of protein energy wasting in chronic kidney disease patients: a consensus statement by the International Society of Renal Nutrition and Metabolism. Kidney Int. 2013 Dec;84(6):1096-107. doi: 10.1038/ki.2013.147. Epub 2013 May 22. PMID 23698226
- [Background] Isoyama N, Qureshi AR, Avesani CM, Lindholm B, Barany P, Heimburger O, Cederholm T, Stenvinkel P, Carrero JJ. Comparative associations of muscle mass and muscle strength with mortality in dialysis patients. Clin J Am Soc Nephrol. 2014 Oct 7;9(10):1720-8. doi: 10.2215/CJN.10261013. Epub 2014 Jul 29. PMID 25074839
- [Background] Chertow GM, Lowrie EG, Wilmore DW, Gonzalez J, Lew NL, Ling J, Leboff MS, Gottlieb MN, Huang W, Zebrowski B, et al. Nutritional assessment with bioelectrical impedance analysis in maintenance hemodialysis patients. J Am Soc Nephrol. 1995 Jul;6(1):75-81. doi: 10.1681/ASN.V6175. PMID 7579073
- [Background] Kalantar-Zadeh K, Kopple JD, Block G, Humphreys MH. A malnutrition-inflammation score is correlated with morbidity and mortality in maintenance hemodialysis patients. Am J Kidney Dis. 2001 Dec;38(6):1251-63. doi: 10.1053/ajkd.2001.29222. PMID 11728958
- [Background] Kalantar-Zadeh K, Kopple JD, Humphreys MH, Block G. Comparing outcome predictability of markers of malnutrition-inflammation complex syndrome in haemodialysis patients. Nephrol Dial Transplant. 2004 Jun;19(6):1507-19. doi: 10.1093/ndt/gfh143. Epub 2004 Apr 6. PMID 15069177
- [Background] Sohrabi Z, Eftekhari MH, Eskandari MH, Rezaeianzadeh A, Sagheb MM. Malnutrition-inflammation score and quality of life in hemodialysis patients: is there any correlation? Nephrourol Mon. 2015 May 23;7(3):e27445. doi: 10.5812/numonthly.7(3)2015.27445. eCollection 2015 May. PMID 26034747